CLINICAL TRIAL: NCT06654674
Title: Gender Differences in Dietary Patterns and Physical Activity: An Insight With Principal Component Analysis (PCA)
Brief Title: Gender Differences in Dietary Patterns and Physical Activity: A PCA Approach
Acronym: GENDPCA
Status: Completed | Type: Observational
Sponsor: San Raffaele Telematic University (Other)
Responsible Party: Principal Investigator, Mauro Lombardo, Mauro Lombardo, MD, Associate Professor in Dietetics and Clinical Nutrition, San Raffaele Telematic University
Other Study IDs: PCA_Gender_2024; 23/13 (Other: Ethics Committee Approval)
Record Dates: First submitted 2024-10-17; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Diet Surveys; Food Preferences
Keywords: Gender Differences; Dietary Patterns; Physical Activity; Principal Component Analysis (PCA); Body Composition; Metabolic Health
MeSH Terms: conditions — Food Preferences; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Participants: This group consists of 2,509 adult participants recruited from a metabolic health center in Rome, Italy. Data on dietary patterns, physical activity, and body composition were collected and analyzed using Principal Component Analysis (PCA) to identify trends and patterns related to gender differences in eating behaviors and physical activity. No specific intervention was applied, as this is an observational study.

SUMMARY:
This study investigates gender differences in dietary patterns and physical activity using Principal Component Analysis (PCA). It aims to identify distinct eating and activity behaviors between men and women in order to develop gender-specific interventions that promote better metabolic health. The study was conducted at a metabolic health center in Rome, Italy, with 2,509 participants. Data were collected through questionnaires and body composition assessments, and PCA was applied to classify participants into groups based on their behaviors.

DETAILED DESCRIPTION:
The study was designed as a cross-sectional analysis of gender differences in dietary patterns and physical activity, utilizing Principal Component Analysis (PCA) to identify distinct behavioral groups. A total of 2,509 participants were recruited from a metabolic health center in Rome, Italy, between May 2023 and June 2024. The study collected detailed data on eating habits, physical activity, and body composition through questionnaires and bioimpedance analysis. Five distinct behavioral groups were identified through PCA, with significant differences in dietary patterns and physical activity levels between men and women. Men were found to consume more meat and participate in strength training, while women favored vegetable-rich diets and had more structured eating routines. These differences also translated into body composition, with men having more lean mass and women more fat mass.

The study highlights the importance of gender-specific interventions in nutrition and physical activity to improve metabolic health outcomes. The results suggest that men could benefit from increased vegetable consumption, while women could benefit from engaging in more physical activity, particularly strength training. Future research should explore these patterns longitudinally to better understand how these behaviors evolve over time and to develop more tailored interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Participants attending the metabolic health center in Rome, Italy.
* Participants who provided informed consent.
* Participants with complete data on dietary patterns, physical activity, and body composition.

Exclusion Criteria:

* Individuals under 18 years of age.
* Participants with diagnosed psychiatric disorders.
* Pregnant women.
* Participants with incomplete or inconsistent data.
* Individuals with alcohol dependence.
* Participants with significant medical conditions that could affect dietary or physical activity assessments (e.g., severe chronic illnesses).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of 2,509 adults attending a metabolic health center in Rome, Italy. These participants were recruited between May 2023 and June 2024. The sample includes both men and women, with a focus on identifying gender-specific patterns in dietary behaviors, physical activity, and body composition. Participants underwent bioimpedance analysis and completed questionnaires regarding their eating habits and physical activity levels.
Sampling Method: Non-Probability Sample
Enrollment: 2509 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Principal Component Analysis (PCA) | Cross-sectional assessment at baseline
  The primary outcome is the identification of distinct dietary patterns and physical activity behaviors based on gender differences.

SECONDARY OUTCOMES:
Physical activity levels based on gender differences | Cross-sectional assessment at baseline
  The study will evaluate how gender differences in physical activity are distributed across different PCA-identified groups

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Caprio, MD, PhD, Study Chair — IRCCS San Raffaele Roma
Locations (1):
- San Raffaele Open University, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be made available to researchers upon reasonable request, provided they submit an appropriate justification for its use.

REFERENCES:
- [Background] Alosaimi N, Sherar LB, Griffiths P, Pearson N. Clustering of diet, physical activity and sedentary behaviour and related physical and mental health outcomes: a systematic review. BMC Public Health. 2023 Aug 18;23(1):1572. doi: 10.1186/s12889-023-16372-6. PMID 37596591
- [Derived] Feraco A, Gorini S, Camajani E, Filardi T, Karav S, Cava E, Strollo R, Padua E, Caprio M, Armani A, Lombardo M. Gender differences in dietary patterns and physical activity: an insight with principal component analysis (PCA). J Transl Med. 2024 Dec 18;22(1):1112. doi: 10.1186/s12967-024-05965-3. PMID 39696430
- [Derived] Feraco A, Armani A, Gorini S, Camajani E, Quattrini C, Filardi T, Karav S, Strollo R, Caprio M, Lombardo M. Gender Differences in Dietary Patterns and Eating Behaviours in Individuals with Obesity. Nutrients. 2024 Dec 6;16(23):4226. doi: 10.3390/nu16234226. PMID 39683619